CLINICAL TRIAL: NCT00222274
Title: A Pilot Study of the Efficacy of Biofeedback in Patients With Fibromyalgia Syndrome.
Brief Title: HRV Biofeedback in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4145
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Fibromyalgia Syndrome
Keywords: fibromyalgia; pain; biofeedback; heart rate variability
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): RSA Biofeedback: RSA Biofeedback Condition. The biofeedback will consist of 10 weekly sessions of training, at the same time of day for each subject. The details of the procedure for RSA biofeedback are described in Appendix A. One single practitioner, a certified biofeedback technician, will provide the biofeedback following the aforementioned protocol. In each session, 20 minutes of biofeedback will be delivered using a J&J C-2+ Physiograph. The participant will be taught to breathe at her resonant frequency, as a first step to training the individual how to produce maximal increases in amplitude of RSA.
  Interventions: Behavioral: RSA Biofeedback
- 2 (Active Comparator): EEG Biofeedback Condition. Participants assigned to this condition will receive 10 sessions of EEG alpha biofeedback. In each session, 20 minutes of biofeedback will be delivered using a J&J I-330-C2+ physiograph. The participant will learn how to modify specific brainwave activity known as alpha. In particular, participants will be taught to increase amplitude of alpha in the range of 8-12 Hz. Increased amplitude is this range is associated with relaxation and reduction of anxiety, but not baroreflex gain. Participants will also practice for two 20-minute periods daily using the same methods used to increase alpha found in lab sessions.
  Interventions: Behavioral: EEG Biofeedback Condition

INTERVENTIONS:
Behavioral: RSA Biofeedback — RSA Biofeedback Condition. The biofeedback will consist of 10 weekly sessions of training, at the same time of day for each subject. The details of the procedure for RSA biofeedback are described in Appendix A. One single practitioner, a certified biofeedback technician, will provide the biofeedback following the aforementioned protocol. In each session, 20 minutes of biofeedback will be delivered using a J&J C-2+ Physiograph. The participant will be taught to breathe at her resonant frequency, as a first step to training the individual how to produce maximal increases in amplitude of RSA.
  Arms: 1
Behavioral: EEG Biofeedback Condition — EEG Biofeedback Condition. Participants assigned to this condition will receive 10 sessions of EEG alpha biofeedback. In each session, 20 minutes of biofeedback will be delivered using a J&J I-330-C2+ physiograph. The participant will learn how to modify specific brainwave activity known as alpha. In particular, participants will be taught to increase amplitude of alpha in the range of 8-12 Hz. Increased amplitude is this range is associated with relaxation and reduction of anxiety, but not baroreflex gain. Participants will also practice for two 20-minute periods daily using the same methods used to increase alpha found in lab sessions.
  Arms: 2

SUMMARY:
A growing body of evidence suggests that the symptoms of many fibromyalgia syndrome (FMS) sufferers might be the result of an imbalance in one of the major stress response systems, the autonomic nervous system. Thus respiratory sinus arrhythmia (RSA) biofeedback, which has shown promise in other conditions associated with an autonomic nervous system imbalance, could be effective in FMS. With the aid of sensors and computers, biofeedback involves modifying and/or learning how to control normally involuntary processes like blood pressure, heart rate and the autonomic nervous system through relaxation and breathing. The goal of this study is to test the effectiveness of a 10-session RSA biofeedback treatment for the symptoms of fibromyalgia. Forty patients receiving the RSA biofeedback treatment will be compared to 40 patients receiving another form of biofeedback thought to be minimally helpful (control group). Later, control group patients will also receive the RSA biofeedback treatment. We will study improvement in symptoms like pain, fatigue, sleep disturbance and depression in the RSA biofeedback group and compare these improvements to those in the control group. We will also assess whether these improvements persist over time and what if any changes in the autonomic nervous system result from the treatment.

DETAILED DESCRIPTION:
Eighty female patients between the ages of 18 and 65 will be recruited from the rheumatology clinic at the University of Medicine and Dentistry of New Jersey - Robert Wood Johnson Medical School (UMDNJ-RWJMS). Qualified participants are those who have a diagnosis of FMS from a board certified rheumatologist using the diagnostic criteria established by the American College of Rheumatology. Because women account for over 85% of FMS patients only women will be included as subjects. Excluded from participating will be women with any of the following medical conditions: neurologic disease or brain injury, stroke or cardiovascular disease, serious pulmonary disease including asthma, liver or kidney disease, serious gastrointestinal disorders, and major psychiatric conditions including psychoses, bipolar disorder, alcohol or drug abuse, and eating disorders. Also excluded will be women with a life threatening medical illness, communicative disorder, lack of fluency in English, illiteracy, cardiac arrhythmia or high frequency and low frequency waves that are indistinguishable or that interact. Patients will be required to add no medications to their regimen during the study period (approximately 5 to 7 months). Based on the clinical judgment of the investigators, patients may also be asked to withdraw from the study should they miss two or more consecutive biofeedback sessions.

After reading and signing the informed consent, all participants will receive a medical evaluation to confirm the diagnosis of FMS based on the criteria established by the American College of Rheumatology. All participants will be evaluated by board certified rheumatologists affiliated with UMDNJ-Robert Wood Johnson Medical School and remain blind to participants' group assignment. This examination will include a baseline tender point count or TPI that will be used as an exploratory measure. Next, participants will be asked to return for an appointment at the Biofeedback Laboratory at UMDNJ-RWJMS. Participants will be instructed to refrain from taking any caffeine or alcohol for twelve hours prior to this and all other sessions where physiologic measures are to be collected. Before beginning physiologic measures assessment, participants will complete the baseline outcome measures, the Fibromyalgia Impact Questionnaire (FIQ), the McGill Pain Questionnaire (MPQ), the Pittsburgh Sleep Quality Inventory (PSQI), and the Beck Depression Inventory II (BDI-II) in a quiet, private room.

The first appointment at the Biofeedback Laboratory will consist of introducing the participant to the setting, equipment and basic procedure of biofeedback. To obtain baseline physiological measures, we will take a 5-minute heart period recording and the other measures including blood pressure, respiration, and muscle tension. For consistency across participants on all resting 5-minute heart period recordings, a "vanilla" baseline task will be included. The "vanilla" baseline is a minimally demanding color detection task shown to provide a stable baseline against which changes in response to experimental challenges can be measured. The task involves the presentation of a 10 to 12 cm rectangle on a computer monitor that changes color every 10 seconds. Six colors are presented randomly and with equal probability over the course of the baseline period. Subjects are told beforehand to count the number of times the object changes back to a randomly determined initial color. At the end of the task subjects are asked to report their count.

All participants will also undergo a simple task for the assessment of orthostatic hypotension. Orthostatic hypotension is defined as a decrease of at least 20 mmHg in systolic blood pressure when an individual moves from a supine to standing position. This assessment will occur in the same lab where the biofeedback session occurs. First, both blood pressure and pulse will be recorded with the participant in a standing position. This will serve as the first recording of BP and pulse measures. Then, the participant will be instructed to lie down completely flat on a floor mat (supine position) for 10 minutes. Approximately three minutes after the participant goes from a supine to standing position, both blood pressure and pulse will be once again recorded. A stand-alone blood pressure device will be used to record these measures.

Next using biofeedback, all participants will be taught to breathe at their resonant frequency as described below. Based on the literature, we will consider the rate of breathing that produces the highest frequency peak to be the participant's "resonant frequency." Finding the true resonant frequency is a complex task beyond the scope and resources of this pilot project. Results from this analysis will advise matching participants on high frequency/low frequency rates.

Group Assignment. Participants will then be randomly assigned to the active treatment group or EEG biofeedback control group using a restricted randomization procedure controlling for age, high frequency/low frequency rates, and general health status. Those assigned to the active treatment group will be given ten weekly training sessions in RSA biofeedback, while those in the control group will receive ten weekly sessions of EEG biofeedback starting immediately. All questionnaire and psychophysiological data collected at baseline will be repeated after the last training session 10 weeks later, and at 3 months. At the end of ten weeks, the EEG biofeedback control group participants will be offered the opportunity to participate in the 10-session RSA biofeedback program and subsequent intervention-related assessments (after the last biofeedback session (10th) and at (3 months). The Week 10 assessment, taken at the conclusion of the EEG biofeedback treatment, will serve as the control group's baseline to maintain 10-week pretest/posttest consistency between groups. EEG biofeedback subjects will be compensated only once if they choose to participate in the RSA biofeedback trial.

EEG Biofeedback Condition. Participants assigned to this condition will receive 10 sessions of EEG alpha biofeedback. In each session, 20 minutes of biofeedback will be delivered using a J&J I-330-C2+ physiograph. The participant will learn how to modify specific brainwave activity known as alpha. In particular, participants will be taught to increase amplitude of alpha in the range of 8-12 Hz. Increased amplitude is this range is associated with relaxation and reduction of anxiety, but not baroreflex gain. Participants will also practice for two 20-minute periods daily using the same methods used to increase alpha found in lab sessions.

RSA Biofeedback Condition. The biofeedback will consist of 10 weekly sessions of training, at the same time of day for each subject. The details of the procedure for RSA biofeedback are described in Appendix A. One single practitioner, a certified biofeedback technician, will provide the biofeedback following the aforementioned protocol. In each session, 20 minutes of biofeedback will be delivered using a J&J C-2+ Physiograph. The participant will be taught to breathe at her resonant frequency, as a first step to training the individual how to produce maximal increases in amplitude of RSA. During the first session, we will measure heart rate oscillation amplitudes while the individual breathes for intervals of two minutes each at specific frequencies, ranging between 4 and 7 breaths per minute, respectively 4, 4.5, 5, 5.5, 6, 6.5, and 7 breaths per minute. We will provide a "pacing stimulus" for this purpose: a light display that moves up and down on the computer screen at the target respiratory rate. The participant will be instructed to breathe at the rate of that stimulus. We will consider the frequency yielding the highest frequency peak on the moving Fourier analysis data collected and displayed by the C-2 physiograph to be the resonant frequency. In subsequent sessions, the individual will be given biofeedback for 20 minutes. The participant will be instructed to practice breathing at her own resonant frequency for 20-minute periods twice daily for the next week. Throughout training the individual will be cautioned to breathe shallowly and naturally, in order to avoid hyperventilation.

At the second session, the participant will be directly given biofeedback for cardiac variability, and instructed to increase the amplitude of heart rate fluctuations that occur in conjunction with respiration. The feedback will be given in several forms. One is using a beat-to-beat cardiotachometer display, superimposed on a measure of respiratory activity taken from a strain gauge. The participant will be instructed to breathe approximately in phase with heart rate changes, with the goal of maximally increasing amplitude of RSA. In another display, the participant will be shown a moving frequency analysis of heart rate, within the band of .005-.4 Hz. The display will be updated approximately every second, and reflects the frequency of heart rate fluctuations within the past 30 seconds. The participant will be instructed to increase the spectral power peak that occurred at approximately resonant frequency. At the beginning and end of this and every biofeedback session participants will be asked to rate their pain, muscle stiffness, fatigue, mood and cognitive processes (memory and concentration) on a verbal scale of one to ten.

In the third session, a stand-alone device will be provided for home practice HeartMath Freeze Framer. This system analyzes heart rhythms and provides a display sensitive to changes. A colorful game format is used to reward the user for increases in heart rate coherence, which in turn will maximize amplitude of RSA. Participants will be instructed to practice for two 20-minute sessions per day and note in the log included with the HeartMath Freeze Framer instructions whether or not they practiced each day, the length of each practice session, and any questions or observations.

Biofeedback Data Collection Procedure. At sessions 1, 10, and at 3 months, a resting 5-minute heart period using the "vanilla" task will be obtained before commencing biofeedback and at the end of the session. During biofeedback, two 5-minute heart period recordings will be taken, one at the beginning of the session and one at the end. Questionnaire data will then be collected. Patients will be given a $25 payment for participation at the end of each data collection session for a total of $75.

ELIGIBILITY:
Inclusion Criteria:

* Qualified participants are those who have a diagnosis of FMS from a board certified rheumatologist using the diagnostic criteria established by the American College of Rheumatology. Because women account for over 85% of FMS patients only women between the ages of 18 and 65 will be included as subjects

Exclusion Criteria:

* Excluded from participating will be women with any of the following medical conditions: neurologic disease or brain injury, stroke or cardiovascular disease, serious pulmonary disease including asthma, liver or kidney disease, serious gastrointestinal disorders, and major psychiatric conditions including psychoses, bipolar disorder, alcohol or drug abuse, and eating disorders. Also excluded will be women with a life threatening medical illness, communicative disorder, lack of fluency in English, illiteracy, cardiac arrhythmia or high frequency and low frequency waves that are indistinguishable or that interact.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Global functioning | 10 weeks

SECONDARY OUTCOMES:
Pain | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Afton L Hassett, Psy.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States